CLINICAL TRIAL: NCT02669121
Title: Phase 2b, Double-Blind, Randomized, Placebo-Controlled Trial to Evaluate the Efficacy and Immunogenicity of the Intramuscular Norovirus GI.1/GII.4 Bivalent Virus-like Particle Vaccine in Healthy Adults Aged 18 - 49 Years
Brief Title: Efficacy and Immunogenicity of Norovirus GI.1/GII.4 Bivalent Virus-like Particle Vaccine in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NOR-211; U1111-1175-9077 (Registry Identifier: WHO)
Record Dates: First submitted 2016-01-27; First posted 2016-01-29 (Estimated); Results first posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Healthy Volunteers
Keywords: Drug therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): NoV placebo-matching 0.5 mL solution for injection, intramuscularly (IM), once, on Day 1.
  Interventions: Biological: NoV Placebo-matching Saline
- NoV GI.1/GII.4 Bivalent VLP Vaccine (Experimental): NoV GI.1/GII.4 bivalent virus-like particle (VLP) vaccine, 0.5 mL injection, intramuscularly (IM), once, on Day 1.
  Interventions: Biological: NoV GI.1/GII.4 Bivalent VLP Vaccine

INTERVENTIONS:
Biological: NoV Placebo-matching Saline — NoV placebo-matching saline (0.9% sodium chloride).
  Arms: Placebo
Biological: NoV GI.1/GII.4 Bivalent VLP Vaccine — NoV bivalent VLP vaccine, adjuvanted with 500 µg aluminum as Al(OH)3.
  Arms: NoV GI.1/GII.4 Bivalent VLP Vaccine

SUMMARY:
The purpose of this study is to evaluate the efficacy of the Norovirus (NoV) GI.1/GII.4 bivalent virus-like particle vaccine against moderate or severe acute gastroenteritis (AGE) due to genotype-specific (GI.1 and GII.4) NoV strains.

DETAILED DESCRIPTION:
The vaccine being tested in this study is called NoV GI.1/GII.4 bivalent VLP vaccine adjuvanted with aluminum hydroxide. The norovirus vaccine is being tested to prevent AGE due to genotype-specific (GI.1 and GII.4) norovirus strains in healthy participants recruited from a US military training installation. This study will look at the illness rate of AGE occurring > 7 days after dosing due to genotype-specific (GI.1 or GII.4) NoV strains represented in the vaccine.

The study will enroll between 2800 and 8700 patients. Participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups-which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

* Norovirus GI.1/GII.4 Bivalent VLP Vaccine
* Placebo (dummy inactive solution) - this is a liquid that looks similar to the study drug but has no active ingredient

All participants will receive one dose of study medication on Day 1 administered via intramuscular injection.

This multi-center trial will be conducted in the United States at select military locations. The overall time to participate in this study is up to 45 days for participants in the navy 53 days for participants in the Air Force, and 72 days for participants in the marines. Participants will make multiple visits to the clinic, including a final visit on the last day of study participation (Day 45, 53 or 72) for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Participant signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any trial procedures after the nature of the trial has been explained according to local regulatory requirements.
2. Male or female participants, 18 to 49 years of age.
3. Is in good health at the time of entry into the trial as determined by medical history and the clinical judgment of the investigator.
4. Can comply with trial procedures and are available for the duration of follow-up.

Exclusion Criteria:

1. Pregnancy.
2. Has known hypersensitivity to any of the Norovirus (NoV) GI.1/GII.4 bivalent virus-like particle (VLP) vaccine components (including excipients).
3. Has known hypersensitivity or allergy to any of the licensed required concomitant vaccine components to be administered (including excipients of these vaccines).
4. Has any condition or circumstance that the investigator determines would interfere with trial evaluation or interpretation.
5. Has known or suspected impairment or alteration of immune function.
6. Has a history of acute gastroenteritis (AGE) within 14 days of enrollment.
7. Has a history of body temperature of 38.0°C (100.4°F) or higher within 3 days of intended trial vaccination.
8. Has received blood, blood products, and/or plasma derivatives or any parenteral immunoglobulin antibody preparation in the past 3 months.
9. Immunosuppressive therapy within 3 months or systemic (e.g., oral or parenteral) corticosteroid treatment within 60 days prior to investigational trial dose administration.
10. Is participating in any clinical trial with another investigational product 30 days prior to the first trial visit or intending to participate in another clinical trial at any time during the conduct of this trial.
11. Participants who are first-degree relatives of individuals involved in the conduct of the trial.
12. Has any history of progressive or severe neurologic disorder, seizure disorder or neuro-inflammatory disease (e.g. Guillain-Barré syndrome).
13. Has history or any illness that, in the opinion of the investigator, might interfere with the results of the trial or pose additional risk to the participants due to participation in the trial.
14. Has received any other vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to enrollment in this trial with the exception of routine immunizations as per Military Procedures.
15. If female of childbearing potential, sexually active, and has not used any of the "acceptable contraceptive methods" for at least 2 months prior to trial entry:

    1. Of childbearing potential is defined as status post onset of menarche and not meeting any of the following conditions: menopausal for at least 2 years, status after bilateral tubal ligation for at least 1 year, status after bilateral oophorectomy, or status after hysterectomy.
    2. Acceptable birth control methods are defined as one or more of the following:

       * Hormonal contraceptive (such as oral, injection, transdermal patch, implant, cervical ring).
       * Barrier (condom with spermicide or diaphragm with spermicide) each and every time during intercourse.
       * Intrauterine device (IUD).
       * Monogamous relationship with vasectomized partner. Partner must have been vasectomized for at least six months prior to the participants' trial entry.
16. If female of childbearing potential and sexually active, refusal to use an "acceptable contraceptive method" from Day 1 through 6 months after the last dose of trial vaccine. In addition, they must be advised not to donate ova during this period.
17. Has any positive or indeterminate pregnancy test.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4748 (Actual)
Dates: Start 2016-06-14 (Actual); Primary Completion 2018-06-16 (Actual); Study Completion 2018-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Great Lakes Naval Station, Great Lakes, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at a single investigative site in the United States from 14 June 2016 to 16 June 2018.
Pre-assignment Details: Healthy volunteers were enrolled in the study and randomized in 1:1 ratio to receive Norovirus GI.1/GII.4 Bivalent VLP Vaccine or Placebo.
Period: Overall Study
Arm/Group | Placebo | NoV GI.1/GII.4 Bivalent VLP Vaccine
Started | 2377 | 2371
Treated (Safety Analysis Set) (All participants who received trial vaccination (NoV or placebo).) | 2357 | 2355
Completed | 2087 | 2089
Not Completed | 290 | 282
Not completed — Adverse Event | 4 | 5
Not completed — Lost to Follow-up | 15 | 27
Not completed — Withdrawal by Subject | 132 | 140
Not completed — Pregnancy | 0 | 1
Not completed — Discharged from US Military Active Service | 117 | 91
Not completed — Reason not Specified | 22 | 18

BASELINE CHARACTERISTICS:
Population: Randomized Set included all enrolled participants.
Groups:
- Placebo: NoV placebo-matching 0.5 mL solution for injection, IM, once, on Day 1.
- NoV GI.1/GII.4 Bivalent VLP Vaccine: NoV GI.1/GII.4 bivalent VLP vaccine, 0.5 mL injection, IM, once, on Day 1.
- Total: Total of all reporting groups
Arm/Group | Placebo | NoV GI.1/GII.4 Bivalent VLP Vaccine | Total
Number analyzed (Participants) | 2377 | 2371 | 4748
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.3 (2.95) | 20.2 (2.74) | 20.3 (2.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 423 | 437 | 860
  Male | 1954 | 1934 | 3888
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 521 | 484 | 1005
  Not Hispanic or Latino | 1856 | 1887 | 3743
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 29 | 27 | 56
  Asian | 87 | 88 | 175
  Native Hawaiian or Other Pacific Islander | 22 | 27 | 49
  Black or African American | 351 | 355 | 706
  White | 1668 | 1667 | 3335
  More than one race | 165 | 146 | 311
  Unknown or Not Reported | 55 | 61 | 116
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2377 | 2371 | 4748

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Moderate or Severe Acute Gastroenteritis (AGE) Occurring for >7 Days After Dosing Due to GI.1 or GII.4 Norovirus Strains (Excluding Co-infection)
Description: Acute gastroenteritis (AGE) is a sudden inflammation or swelling in the lining of the stomach causing diarrhea and vomiting. A norovirus AGE case was defined as meeting the work-up definition plus a norovirus positive stool sample or vomitus sample confirmed by reverse transcriptase polymerase chain reaction (RT-PCR). The severity of AGE was graded by the investigator as per CTCAE criteria. AGE occurring due to NoV strains excluding co-infection with Salmonella, Shigella or Campylobacter is reported. The Norovirus strains included: GI.1, GI.7a, GII.2 and GII.4.
Time Frame: Up to Day 47
Population: Full Analysis Set included all participants who were randomized and received the trial dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | NoV GI.1/GII.4 Bivalent VLP Vaccine
Number analyzed (Participants) | 2357 | 2355
Participants | 5 | 1
Statistical Analysis 1: Comparison: Placebo vs NoV GI.1/GII.4 Bivalent VLP Vaccine; Test type: Superiority; Cox Proportional Hazard = 0.800, 99.99% CI 2-sided [-13.181 to 0.997]; The vaccine efficacy was met if lower bound of confidence interval (CI) for vaccine efficacy was above 0. Vaccine efficacy (VE) was defined as 1-(hazard rate for NoV vaccine arm / hazard rate for placebo arm), where the hazard ratio is from the Cox proportional hazard (PH) model. The 99.99% CI for the VE was obtained by taking 1 minus the 99.99% CI of the hazard ratio from the PH model

2. Secondary Outcome: Number of Participants With Moderate or Severe AGE Occurring >7 Days After Dosing Due to Any Norovirus Strain (Excluding Co-infection)
Description: Acute gastroenteritis (AGE) is a sudden inflammation or swelling in the lining of the stomach causing diarrhea and vomiting. A norovirus AGE case was defined as meeting the work-up definition plus a norovirus positive stool sample or vomitus sample confirmed by RT-PCR. The severity of AGE was graded by the investigator as per CTCAE criteria. AGE occurring due to NoV strains excluding co-infection with Salmonella, Shigella or Campylobacter is reported. The Norovirus strains included: GI.1, GI.7a, GII.2 and GII.4.
Time Frame: Up to Day 47
Population: Full Analysis Set included all participants who were randomized and received the trial dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | NoV GI.1/GII.4 Bivalent VLP Vaccine
Number analyzed (Participants) | 2357 | 2355
Participants | 26 | 10
Statistical Analysis 1: Comparison: Placebo vs NoV GI.1/GII.4 Bivalent VLP Vaccine; Test type: Superiority; Cox Proportional Hazard = 0.618, 95.01% CI 2-sided [0.208 to 0.816]; The vaccine efficacy was met if lower bound of CI for vaccine efficacy was above 0. Vaccine efficacy (VE) was defined as 1-(hazard rate for NoV vaccine arm / hazard rate for placebo arm), where the hazard ratio is from the PH model. The 95.01% CI for the VE was obtained by taking 1 minus the 95.01% CI of the hazard ratio from the PH model

3. Secondary Outcome: Number of Participants With Moderate or Severe AGE Occurring >7 Days After Dosing Due to Any Norovirus Strain (Including Co-infection)
Description: Acute gastroenteritis (AGE) is a sudden inflammation or swelling in the lining of the stomach causing diarrhea and vomiting. A norovirus AGE case was defined as meeting the work-up definition plus a norovirus positive stool sample or vomitus sample confirmed by RT-PCR. The severity of AGE was graded by the investigator as per CTCAE criteria. AGE occurring due to NoV strains including co-infection with Salmonella, Shigella or Campylobacter is reported. The Norovirus strains included: GI.1, GI.7a, GII.2 and GII.4.
Time Frame: Up to Day 47
Population: Full Analysis Set included all participants who were randomized and received the trial dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | NoV GI.1/GII.4 Bivalent VLP Vaccine
Number analyzed (Participants) | 2357 | 2355
Participants | 26 | 10
Statistical Analysis 1: Comparison: Placebo vs NoV GI.1/GII.4 Bivalent VLP Vaccine; Test type: Superiority; Cox Proportional Hazard = 0.618, 95% CI 2-sided [0.208 to 0.816]; The vaccine efficacy was met if lower bound of CI for vaccine efficacy was above 0. Vaccine efficacy (VE) was defined as 1-(hazard rate for NoV vaccine arm / hazard rate for placebo arm), where the hazard ratio is from the PH model. The 95% CI for the VE was obtained by taking 1 minus the 95% CI of the hazard ratio from the PH model

4. Secondary Outcome: Number of Participants With Moderate or Severe AGE Occurring >7 Days After Dosing Due to GI.1 or GII.4 Norovirus Strains (Including Co-infection)
Description: as for outcome 3
Time Frame: Up to Day 47
Population: Full Analysis Set included all participants who were randomized and received the trial dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | NoV GI.1/GII.4 Bivalent VLP Vaccine
Number analyzed (Participants) | 2357 | 2355
Participants | 5 | 1
Statistical Analysis 1: Comparison: Placebo vs NoV GI.1/GII.4 Bivalent VLP Vaccine; Test type: Superiority; Cox Proportional Hazard = 0.800, 95% CI 2-sided [-0.711 to 0.977]; [other analysis details as in outcome 3, analysis 1]

ADVERSE EVENTS:
Time Frame: From Day 1 up to the end of the study (Up to 47 days)
Description: At each visit investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by participant or observed by investigator was recorded, irrespective of relation to study treatment. Safety Analysis Set included all participants who received trial dose (NoV GI.1/GII.4 bivalent VLP vaccine or saline placebo).
Arm/Group | Placebo | NoV GI.1/GII.4 Bivalent VLP Vaccine
All-Cause Mortality (participants affected / at risk) | 0/2357 | 0/2355
Serious Adverse Events (participants affected / at risk) | 35/2357 | 29/2355
Other Adverse Events (participants affected / at risk) | 88/2357 | 98/2355
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=2357) | NoV GI.1/GII.4 Bivalent VLP Vaccine (N=2355)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 2
Gastroenteritis (Infections and infestations) | 1 | 2
Cellulitis staphylococcal (Infections and infestations) | 0 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 2
Infectious mononucleosis (Infections and infestations) | 2 | 0
Subcutaneous abscess (Infections and infestations) | 2 | 0
Abscess jaw (Infections and infestations) | 1 | 0
Abscess oral (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Chlamydial infection (Infections and infestations) | 1 | 0
Gastroenteritis clostridial (Infections and infestations) | 0 | 1
Helicobacter gastritis (Infections and infestations) | 1 | 0
Helicobacter infection (Infections and infestations) | 0 | 1
Parotitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Staphylococcal abscess (Infections and infestations) | 0 | 1
Tonsillitis streptococcal (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Varicella (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 | 3
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Myelopathy (Nervous system disorders) | 1 | 0
Adjustment disorder (Psychiatric disorders) | 5 | 2
Adjustment disorder with depressed mood (Psychiatric disorders) | 1 | 3
Depressed mood (Psychiatric disorders) | 0 | 2
Major depression (Psychiatric disorders) | 1 | 1
Persistent depressive disorder (Psychiatric disorders) | 1 | 1
Suicidal ideation (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 0 | 1
Panic attack (Psychiatric disorders) | 1 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=2357) | NoV GI.1/GII.4 Bivalent VLP Vaccine (N=2355)
Upper respiratory tract infection (Infections and infestations) | 45 | 57
Procedural pain (Injury, poisoning and procedural complications) | 57 | 55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/21/NCT02669121/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-14): https://cdn.clinicaltrials.gov/large-docs/21/NCT02669121/SAP_001.pdf